CLINICAL TRIAL: NCT04166825
Title: The Impact of Different Ovarian Hyperstimulation Protocols on Coagulation and Fibrinolysis.
Brief Title: Ovarian Hyperstimulation and Fibrin Clot Properties.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Magdalena Piróg, MD, Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 292/B/2014/MP
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Fibrin Blood Clot; Infertility, Female; Endometriosis
Keywords: coagulation; fibrinolysis; ovarian hyperstimulation; infertility
MeSH Terms: conditions — Infertility, Female; Endometriosis; Thrombosis; Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Long protocol (Active Comparator): Ovarian hyperstimulation started on day 2 or 3 of the cycle with daily subcutaneous injections of recombinant human FSH (follitropin α, Gonal F®, Merck Serono) and/or urinary human menopausal gonadotropin (menotropin, Menopur®, Ferring GmbH) or mixed recombinant human FSH/LH (Pergoveris®, Merck Serono) with a starting dose of 87.5-250 IE/day
  Interventions: Diagnostic Test: fibrin clot properties
- Short protocol (Active Comparator): Ovarian hyperstimulation with a GnRH-antagonist consisted of the use of ganirelix (Orgalutran®, MSD) from the 6th day of stimulation until it's end at the daily dose of 0.25 mg
  Interventions: Diagnostic Test: fibrin clot properties
- Clomiphene citrate (Active Comparator): Ovarian stimulation with clomiphene citrate (Clostilbegyt®, EGIS) 50 mg daily per os form 3rd to 7th day of the cycle
  Interventions: Diagnostic Test: fibrin clot properties
- Letrozole (Active Comparator): Ovarian stimulation with letrozole (Lametta®, Vipharm) 2.5 mg daily per os form 3rd to 7th day of the cycle
  Interventions: Diagnostic Test: fibrin clot properties
- Gonadotropins (Active Comparator): Ovarian hyperstimulation started on day 2 or 3 of the cycle with daily subcutaneous injections of recombinant human FSH (follitropin α, Gonal F®, Merck Serono).
  Interventions: Diagnostic Test: fibrin clot properties

INTERVENTIONS:
Diagnostic Test: fibrin clot properties — Assessment of thrombin generation and efficiency of fibrinolysis.

SUMMARY:
The impact evaluation of ovarian hyperstimulation on coagulation and fibrinolysis in infertile women.

Comparative analysis between different ovarian stimulation protocols on thrombin formation and efficiency of fibrinolysis in women diagnosed with infertility.

DETAILED DESCRIPTION:
Infertility is a common problem. Assisted reproductive techniques (ART) increases the chance of getting pregnant by couples undergoing such treatment. Unfortunately, the numer of live births after ART remains still low. Over the past three decades, physicians have tried to improve infertility diagnosis and increase its successful treatment. An effort aimed at increasing effectivenes of diagnosis resulted in hypothesis that one of probable reasons of infertility may be the occurrence of microclots, which worsen implantation and embryos development. There are currently no published studies describing the effects of different ovarian hyperstimulation protocols on hemostasis (coagulation and fibrinolysis).

The parameters of thrombin generation and efficiency of fibrinolysis will be evaluated in women qualified for ovarian hyperstimulation. The study may improve the effectiveness of ART.

ELIGIBILITY:
Inclusion Criteria:

* infertility defined based on the WHO 2010 criteria

Exclusion Criteria:

* ovarian involvement
* oral contraceptives use within previous 3 months
* dienogest therapy within 3 months until ART
* thrombotic events in the medical history
* severe hypertension
* diabetes mellitus
* the presence of known VTE risk factors, including obesity, recent major surgery with prolonged immobilization or trauma,
* deficiency of antithrombin, protein C or protein S,
* antiphospholipid syndrome,
* known malignancy,
* any chronic inflammatory diseases (e.g. rheumatoid arthritis)
* advanced chronic renal disease (estimated glomerular filtration rate [eGFR] <30 ml/min),
* international normalized ratio (INR) more than 1.2 at the day of blood draw
* pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fibrin clot properties before and after the ovarian hyperstimulation. | 4 months
  Coagulation (endogenous thrombin potential) and fibrinolysis (F1+2, clot lysis time)parameters assessment.

SECONDARY OUTCOMES:
Endometriosis and fibrin clot properties. | 1 cycle
  Changes of fibrin clot properties before and after ovarian hyperstimulation in women with endometriosis - Coagulation (endogenous thrombin potential) and fibrinolysis (F1+2, clot lysis time)parameters assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecological Endocrinology Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pirog M, Kacalska-Janssen O, Jach R, Wyroba J, Chrostowski B, Zabczyk M, Natorska J. GnRH Antagonist Protocol Enhances Coagulation During Controlled Ovarian Stimulation for IVF. Reprod Sci. 2022 Dec;29(12):3521-3531. doi: 10.1007/s43032-022-01026-6. Epub 2022 Jul 12. PMID 35821349